CLINICAL TRIAL: NCT05462327
Title: Low Fresh Gas Flow and Normal Gas Flow Anesthesia in Patients Undergoing Surgery in Prone Position: Impact on Hemodynamics and Regional Cerebral Oxygenation
Brief Title: Low Fresh Gas Flow in Prone Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Esra Akdaş Tekin, Medical Doctor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 48670771-514.10/1477
Record Dates: First submitted 2022-07-06; First posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Anesthesia
Keywords: Hemodynamics; Low Flow Anesthesia; Near Infrared Spectroscopy; Prone Positioning; Regional Cerebral Oxygenation
MeSH Terms: interventions — Prone Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Fresh Gas Flow in Prone Position (Experimental): Low fresh gas flow (0,5 L/min during maintenance)
  Interventions: Procedure: Low Fresh Gas Flow in Prone Position
- Normal Fresh Gas Flow in Prone Position (Active Comparator): Normal flow (2 L/min) in general anesthesia.
  Interventions: Procedure: Normal Fresh Gas Flow in Prone Position

INTERVENTIONS:
Procedure: Low Fresh Gas Flow in Prone Position — In the low fresh gas flow group, the flow rate was reduced to 0.5 L/min
  Arms: Low Fresh Gas Flow in Prone Position
Procedure: Normal Fresh Gas Flow in Prone Position — In the normal flow rate group, the gas flow rate was reduced to 2 L/min during the maintenance phase.
  Arms: Normal Fresh Gas Flow in Prone Position

SUMMARY:
Low flow anesthesia in the prone position was safe in terms of systemic hemodynamics and did not reduce cerebral oxygenation compared to normal flow.

DETAILED DESCRIPTION:
Patients were randomly allocated to either low fresh gas flow(LF, 0,5 L/min during maintenance) or normal flow (NF, 2 L/min)) general anesthesia. In both groups, participants were first administered with 100% oxygen at a 4 L/min flow rate. Propofol 2-2,5 mg/kg, rocuronium bromide 0,6 mg/kg, and fentanyl 1 mcg/kg IV were used for anesthesia induction.In the operating room, pulse rate, mean arterial pressure (MAP), peripheral hemoglobin oxygen saturation (spO2), and right and left side regional cerebral oxygen saturation (Masimo's O3 regional oximetry device) were measured before premedication and anesthesia induction, at 10 minutes after endotracheal intubation, at 10 minutes after prone positioning, at 1st, 2nd, 3rd, 4th and 5th hours of operation, before repositioning to supine, after the resumption of supine position and at 5 minutes after extubation. In conclusion, low flow anesthesia in patients undergoing surgery in the prone position did not cause a reduction in cerebral oxygenation compared to normal flow.

ELIGIBILITY:
Inclusion Criteria:

* undergoing surgery in the prone position
* having an American Society of Anesthesiologists (ASA) physical status I to III
* willingness to participate in the study

Exclusion Criteria:

* having a Glasgow coma scale (GSC) score ≤ 12
* previous history of cranial surgery
* advanced cardiovascular and/or pulmonary disease
* mental retardation
* neurological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Low and Normal Fresh Gas Flow Difference in Prone Position | Systemic and cerebral oxygenation values were measured 10 minutes after induction to general anesthesia and followed up to 10 minutes were left to completion of the surgery for about 5 hours, which may vary according to the duration of the surgery.
  Whether low flow anesthesia in the prone position is safe in terms of systemic hemodynamics and cerebral oxygenation compared to normal flow anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Tascioglu City Hospital, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Patient's sex, ages and additional conditions